CLINICAL TRIAL: NCT02878694
Title: Treatment of Ptosis to Muscular Dystrophy Oculopharyngeal by Myoblast Autologous Graft
Acronym: TTT-PT-DOP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other); Rennes University Hospital (Other); Centre Hospitalier Universitaire, Amiens (Other); University Hospital, Lille (Other); University Hospital, Brest (Other); Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001192-48
Record Dates: First submitted 2016-03-08; First posted 2016-08-25 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Muscular Dystrophy, Oculopharyngeal; Ptosis
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myoblast autologous graft (Experimental): 30 million autologous myoblasts in 6 intramuscular injections
  Interventions: Biological: Myoblast autologous graft

INTERVENTIONS:
Biological: Myoblast autologous graft — 30 million autologous myoblasts in 6 intramuscular injections No treatment in the second eye

SUMMARY:
Interventional , multicenter , comparative study. One eye receiving the cells and the contralateral eye as a negative control . If effectiveness following review of the primary endpoint and the advice of an independent expert committee , the experimental treatment will be offered to the patient to the contralateral eyelid.

Objective is to restore muscle function levator muscle of the upper eyelid by providing a registry of autologous myoblasts from a non- clinically affected muscle .

DETAILED DESCRIPTION:
Muscular dystrophy oculopharyngeal ( OPMD ) is an autosomal dominant inherited myopathy manifested as selective involvement of the levator muscles of the upper eyelids , head of ptosis, and muscles of the intersection pharyngolaryngeal originally disorders swallowing. Ptosis can be treated with surgery ( shortening of the levator muscle ), but the disease continues to evolve , relapses occur , necessitating another intervention , which is the suspension of the eyelid to the frontal muscle that can cause corneal complications by imperfect lid closure .

Main objective is to restore muscle function levator muscle of the upper eyelid by providing a registry of autologous myoblasts from a non- clinically affected muscle .

A study on the same model was conducted in patients in ENT OPMD crossroads of muscles with encouraging results , 12/12 patients had improved quality of life and no degradation of swallowing was observed in 10 / 12 patients.

This is an interventional study , multicenter, comparative , one eye receiving the cells and the contralateral eye as a negative control . If effectiveness following review of the primary endpoint and the advice of an independent expert committee , the experimental treatment will be offered to the patient to the contralateral eyelid.

Seven centers are associated with this project as inclusion and assessment center. Patients are referred by different clinical sites in Caen ophthalmology department which will be performed pre-transplant assessment, the collection of donor myoblast muscle graft and part tracking.

The expected duration is 3 years (2 years of inclusion and evaluation of the primary endpoint at 1 year) for inclusion of 10 patients.

The safety of autologous myoblast transplantation has been shown in several directions with promising efficacy results. They will be produced by the unit of Biotherapy Rouen University Hospital (Prof. O. Boyer), who currently leads a test with these cells (ClinicalTrials.gov, myoblast for Anal Incontinence (MIAS), NCT01523522, 24 patients were provided in Protocol was included in July 2014, at 6 months follow up of the last patient is expected in January 2015) and authorized the production of advanced therapy medicinal products prepared punctually (ANSM).

In this study, different successive steps:

* Step of including: patient aged 18 to 75, verification of the diagnosis of the disease, evaluation balance ptosis (measurements, photographs, films), obtaining consent,
* Muscle biopsy of a healthy muscle to cell amplification, an outpatient basis, under local anesthesia, 3 to 4 weeks before transplantation,
* Transplant myoblasts by multiple intramuscular injections (6), under local anesthesia. Longitudinal microscarifications be made superficially injected into muscles to stimulate muscle regeneration. Intramuscular injection of myoblasts will be in the levator muscle of the upper lid 6 in equidistant points, each injection containing 5 million cells. These injections will be made in muscle mass over an area of about 5 cm2, ranging between 6 and 20 mm above the tarsus to be in the thick muscle area. It is intended to be injected into the eye to treat randomized a total of 30 million myoblasts. This protocol is based on the one used for correction of ENT disorders within several PHRC under the responsibility of Professor Sophie Périé. The doses used for the myoblast transplantation in the pharyngeal constrictor muscles were adapted to the levator muscle of the eyelid.
* Follow-up visits for 3 years for each patient:

  * The first year, to evaluation of the primary endpoint visit to 8 days to a month, then every 3 months
  * Out protocol and up to 3 years after administration of the cells every 6 months (this monitoring will be carried out as part of standard care).

These visits evaluate the effectiveness of the transplant on different objective measurements on both eyes (eyelid opening slot in the gaze straight ahead; levator muscle strength of the upper eyelid, visual benefit: measurement of visual acuity measurement visual field), and the profit on neck pain. The tours include a side effect detection examination (local inflammatory phenomena, palpable lumps).

In the end, this landmark trial for the new F.H.U. SURFACE dealing with regenerative medicine in the head and neck, the investigators expect an improvement in the quality of the levator of the upper eyelid muscles deficient with a correction of ptosis in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ( with suitable contraception) over 18 years of age 75
* OPMD confirmed by genetic diagnosis ( gene mutation PABPN1 by triplet expansion GCG)
* OPMD with ptosis
* Obtaining informed consent signed

Exclusion Criteria:

* Evolutionary contagious infectious pathology
* Inflammatory diseases
* Any other neuromuscular disease
* Malignant tumor pathology of history
* Renal impairment ( creatinine clearance < 60ml / min)
* Hepatic insufficiency
* Pregnant woman confirmed by a dosing B-HCG or lactating
* Inability to perform a muscle biopsy
* Preparation of myoblasts uncommitted to step 2nd release
* Inability to follow up to 36 months
* Refusal to sign the consent form
* No Social Security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Improvement of ptosis | baseline and 12 months
  The improvement in ptosis is considered by measuring the opening of the lid gap ( OFP) , the gaze straight ahead and no inclination of the head, the eye untreated and treated before and after treatment at 12 month.

SECONDARY OUTCOMES:
acuity | 12 months
  Measure of visual acuity ( without lifting the lid manually and without head tilt ) according Monoyer scale ,
Goldmann Visual Field | 12 months
neck pain with Visual Analaogue Scale | 12 months
Tolerance of the sampling procedure and transplantation, swelling (yes / no) | baseline
Tolerance of the sampling procedure and transplantation : visual analogue scale Pain about the procedure | baseline
Tolerance of collection of the seat and transplantation: hematoma (yes / no ) | baseline
fever | baseline
strength of the levator muscle of the upper eyelid | 12 months
  This is assessed by measuring the travel of the free edge of the upper eyelid between the eyes down and look up blocking the frontal muscle (photos and films) . Normal Range : 15 to 17 mm. Very impaired in patients with DOP .

CONTACTS AND LOCATIONS:
Overall Officials: Françoise CF Chapon, PhD, Study Chair — CHU CAEN; Olivier BO Boyer, PhD, Study Chair — CHU Rouen; Frederic MF Mouriaux, PhD, Study Chair — CHU Rennes; Sophie PS Perie, PhD, Study Chair — APHP
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No